CLINICAL TRIAL: NCT02248155
Title: Sifrol® Onset of Action and Impact on RLS: A 12-week Observational Study in Patients With Primary RLS
Brief Title: Observational Study of Sifrol® in Patients With Primary Restless Legs Syndrome (RLS)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.618
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- RLS patients
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Pramipexole
  Other Names: Sifrol®

SUMMARY:
The objectives of this Post Marketing Surveillance (PMS) are:

* Evaluation of the treatment effect of pramipexole on Restless Legs Syndrome (RLS) severity as measured by International Restless Legs Syndrome Scale (IRLS) and Clinical Global Impression Improvement scale (CGI- I)
* Evaluation of the time to reaching maintenance dose of pramipexole
* Evaluation of work productivity impairment associated with RLS based on the Work Productivity and Activity Impairment Questionnaire (WPAI) questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from primary RLS who are eligible for Pramipexol (PPX) treatment could be included into the study
* Patients not pre-treated with any dopaminergic agent (de novo patients) or patients pre-treated with dopaminergic medication
* Male of female patients of any age

Exclusion Criteria:

* The treating physicians are asked to consider the regulations described in the Summary of Product Characteristics (SmPC) for the treatment with pramipexole

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from moderate to severe RLS recruited at office-based general practitioners and interists
Sampling Method: Non-Probability Sample
Enrollment: 2644 (Actual)
Dates: Start 2006-04; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Assessment of RLS symptoms (IRLS) on a 4-point rating scale | up to 12 weeks
Change from Baseline in WPAI by means of a patient questionnaire | Baseline, 12 weeks

SECONDARY OUTCOMES:
Number of patients with adverse drug reactions | up to 12 weeks
Global assessment of efficacy by investigator on a 5-point scale | after 12 weeks
Change in Clinical Global Impression Improvement (CGI-I) rated on a 7-point scale | up to 12 weeks
Time to reach pramipexol maintenance dose | up to 12 weeks